CLINICAL TRIAL: NCT01642537
Title: Electroanatomical Mapping of Patients Undergoing Catheter Ablation Procedures Using Rhythmia Mapping System and Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TP000-147
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rhythmia Mapping System & Catheter (Other): This is a single arm diagnostic feasibility study with the Rhythmia Mapping System and the Rhythmia Mapping Catheter
  Interventions: Device: Rhythmia Mapping System and the Rhythmia Mapping Catheter

INTERVENTIONS:
Device: Rhythmia Mapping System and the Rhythmia Mapping Catheter — Patients will undergo a diagnostic assessment with the Rhythmia Mapping System and the Rhythmia Mapping Catheter as part of the Electrophysiology Ablation Procedure.

SUMMARY:
The purpose of this study is a feasibility study for the Rhythmia Medical Mapping System and Mapping Catheter on patients undergoing catheter ablation procedures for the treatment of cardiac tachyarrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. Patient understands the implications of participating in the study and provides informed consent
2. Patient is willing to comply with specified follow-up evaluation and can be contacted by telephone
3. Patients referred for a catheter ablation procedure to treat an atrial or ventricular arrhythmia
4. Patient can be heparinized during the procedure

Exclusion Criteria:

1. Patients requiring an emergency ablation procedure
2. Patients hemodynamically unstable
3. Patients with NYHA Class III or IV heart failure
4. Women who are pregnant or lactating
5. Patients having cardiac surgery within the past two months
6. Patients with Long QT Syndrome, Brugada Syndrome, or Torsade de Pointes
7. Patients with intracardiac thrombus, tumor, or other abnormality which precludes catheter introduction
8. Patients with acute myocardial infarction within 3 months
9. Patients awaiting cardiac transplantation
10. Patients enrolled in any other clinical study
11. Patients with an age <18 or >75 years
12. Patients with stable/unstable angina or ongoing myocardial ischemia
13. Patients with congenital heart disease (not including atrial septal defect (ASD) or patent foramen ovale (PFO) without a right to left shunt) where the underlying abnormality increases the risk of an ablative procedure
14. Patients with pulmonary hypertension (mean or systolic pulmonary artery (PA) pressure > 50mm Hg on Doppler echo)
15. Patients with a left atrial diameter > 55 mm
16. Patients with any arrhythmia currently being treated where the arrhythmia or the management may interfere with this study
17. Patients with active infection or sepsis
18. Patients with untreatable allergy to contrast media
19. Patients with a history of blood clotting (bleeding or thrombotic) abnormalities
20. Patients with any known sensitivities to heparin or warfarin
21. Patients with severe chronic obstructive pulmonary disease (COPD) (identified by a forced expiratory volume [FEV1] <1)
22. Patients with severe co morbidity or poor general physical/mental health that, in the opinion of the investigator, will not allow the patient to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life expectance, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Major device related adverse cardiac and cerebrovascular events | 30 days
Device Performance | 1 day- Procedure

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada